CLINICAL TRIAL: NCT07261592
Title: Entinostat Combined With Chemotherapy as Second-line Therapy for Unresectable Locally Advanced or Metastatic Bladder Cancer: A Single-arm, Prospective Clinical Trial
Brief Title: Entinostat & Chemotherapy for Locally Advanced or Metastatic Bladder Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-UC-108
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer; Histone Deacetylase Inhibitor; Entinostat; Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — entinostat; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Entinostat plus chemotherapy (Experimental): The study was divided into two phases: chemotherapy phase and continuous treatment phase. During chemotherapy phase, patients receive 6 cycles of GC (gemcitabine and cisplatin) chemotherapy along with entinostat followed by efficacy evaluation. If stable disease is reached according to RECIST 1.1 criteria, patients may receive continuous entinostat treatment until disease progression or intolerable side effects.
  Interventions: Drug: Entinostat; Drug: Chemotherapy

INTERVENTIONS:
Drug: Entinostat — Take entinostat 5mg orally once weekly (at least 1 hour before meal and 2 hours after meal).
Drug: Chemotherapy — Gisantinib and cisplatin chemotherapy for 6 cycles, 21 days per cycle. Gisantinib 1000mg/m2 is given intravenously on Day 1 and 8 for each cycle while cisplatin 70mg/m2 is given intravenously on Day2.

SUMMARY:
This single-center single-arm, open-label prospective clinical trial aimed to evaluate the efficacy and safety of entinostat combined with chemotherapy as second-line therapy for unresectable locally advanced or metastatic bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic confirmed unresectable advanced or metastatic bladder cancer, except for those with squamous differentiation, glandular differentiation or both;
* Failure of first-line treatment;
* There is at least one measurable lesion according to RECIST 1.1;
* Archived tumor tissue samples or tumor biopsies must be provided;
* ECOG score of 0-1 an an estimated survival of at least 6 months;
* Adequate organ function;
* Patients voluntarily participated in this study, signed the informed consent form, and had good compliance;
* Women with fertility must consent to contraception during the study and for 6 months after the last dose of study drug.

Exclusion Criteria:

* Patients who received platinum-based chemotherapy after failure of first-line treatment;
* Patients who received platinum-based chemotherapy withnin a 24 month before this trial;
* Those who have received other anti-tumor treatment or participated in other clinical studies within 4 weeks before the start of the study, or have not recovered from the last toxicity (except grade 2 hair loss and grade 1 neurotoxicity);
* Concomitant disease such as uncontrolled hypertension or diabetes, renal inadequacy, myocardial infarction, severe angina;
* Female subjects who are pregnant, breastfeeding or planning to become pregnant during the study;
* Patients with serious physical or mental illnesses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | 36 months
  ORR refers to the percentage of confirmed cases of complete response (CR) and partial response (PR) according to the RECIST (Response Evaluation Criteria in Solid Tumours) version 1.1.

SECONDARY OUTCOMES:
ProgressionFree Survival, PFS | 36 months
  PFS refers to the time from the beginning of treatment to disease progression or death from any reason (whichever occurs first).
Overall Survival, OS | 36 months
  OS refers to the time from the beginning of treatment to death from any reason.
Disease Control Rate, DCR | 36 months
  The percentage of cases with CR, PR, and SD (≥4 weeks) among patients with evaluable efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, PhD, Principal Investigator — Nanjing University Medical School Affiliated Nanjing Drum Tower Hospital
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code